CLINICAL TRIAL: NCT00958776
Title: A Phase 3, Multicenter, Randomized, Double-blind, Controlled Study to Evaluate the Efficacy and Safety of Peramivir Administered Intravenously in Addition to Standard of Care Compared to Standard of Care Alone in Adults and Adolescents Who Are Hospitalized Due to Serious Influenza
Brief Title: A Study to Evaluate the Efficacy and Safety of IV Peramivir in Addition to Standard of Care Compared to Standard of Care Alone in Adults and Adolescents Who Are Hospitalized Due to Influenza
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated for futility
Sponsor: BioCryst Pharmaceuticals (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCX1812-301
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-01

CONDITIONS: Cough; Sore Throat; Nasal Congestion; Headache; Fever; Seasonal Influenza
Keywords: Influenza; Hospitalized; Antiviral; Flu
MeSH Terms: conditions — Cough; Pharyngitis; Nasal Obstruction; Headache; Fever; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peramivir+SOC (Experimental): * Adults (≥ 18 years): Peramivir (BCX-1812) 600 mg, administered intravenously, once daily (every 24 hrs) for 5 days (5 doses) in addition to institution's standard of care.
  * Adolescents (12-17 years): Peramivir (BCX-1812) 10 mg/kg (not to exceed a maximum dose of 600 mg), administered intravenously, once daily (every 24 hrs) for 5 days (5 doses) in addition to institution's standard of care.
  Interventions: Drug: Peramivir+SOC
- Placebo+SOC (Placebo Comparator): Placebo Peramivir (BCX1812) administered intravenously, once daily (every 24 hrs) for 5 days (5 doses) in addition to institution's standard of care.
  Interventions: Drug: Placebo+SOC

INTERVENTIONS:
Drug: Peramivir+SOC — * Adults (≥ 18 years): Peramivir (BCX-1812) 600 mg, administered intravenously, once daily (every 24 hrs) for 5 days (5 doses) in addition to institution's standard of care.
  * Adolescents (12-17 years): Peramivir (BCX-1812) 10 mg/kg (not to exceed a maximum dose of 600 mg), administered intravenously, once daily (every 24 hrs) for 5 days (5 doses) in addition to institution's standard of care.
  Arms: Peramivir+SOC
Drug: Placebo+SOC — Placebo Peramivir (BCX1812) administered intravenously, once daily (every 24 hrs) for 5 days (5 doses) in addition to institution's standard of care.
  Arms: Placebo+SOC

SUMMARY:
A Phase 3, multicenter, randomized, double-blind, controlled study to evaluate the efficacy and safety of peramivir administered intravenously in addition to standard of care compared to standard of care alone in adults and adolescents who are hospitalized due to serious influenza.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years of age, male or female.
* Able to provide informed consent, or for whom consent may be provided by guardian, unless informed consent provided by a guardian or a legally authorized representative is not consistent with applicable local or ethical concerns, procedures, directives and/or guidelines.
* Subject must have at least one of the following clinical presentations at Screening:

  1. Oral temperature ≥ 38.0 °C (≥100.4 °F), ≥38.6°C (≥101.4 °F) tympanic or rectal OR
  2. Oxygen saturation <92%, OR
  3. Two out of the following three vital signs:

Respiration rate >24/minute, Heart rate >100/minute, Systolic BP <90 mmHg

* Presence of at least one respiratory symptom (cough, sore throat, or nasal congestion) of any severity (mild, moderate, or severe).
* Presence of at least one constitutional symptom (headache, myalgia, feverishness, or fatigue) of any severity (mild, moderate, or severe).
* Onset of illness no more than 72 hours before presentation. Note: Time of onset of illness is defined as the earlier of either (1) the time when the temperature was first measured as elevated, OR (2) the time when the subject experienced the presence of at least one respiratory symptom AND the presence of at least one constitutional symptom.
* Either:

Severity of illness that, in the Investigator's judgment, justifies hospitalization of the subject for supportive care.

OR

Presence of one or more of the following factors:

Age ≥60 years. Presence of chronic obstructive pulmonary disease (COPD) or other chronic lung disease requiring daily pharmacotherapy.

Current history of congestive heart failure or angina. Presence of diabetes mellitus, clinically stable or unstable. Transcutaneous oxygen saturation <94% without supplemental oxygen for at least 5 minutes, or a medically significant decrease in oxygen saturation from an established baseline value (an investigative site at altitude >2000 ft above sea level will utilize different criteria for oxygen saturation).

History of chronic renal impairment not requiring peritoneal dialysis. Serum creatinine > 2.0 mg/dL or > 177 μmol/L.

* Diagnosis of Influenza by satisfying one of the following:

  1. Clinical Influenza with Positive Diagnostic Test. Subjects who have a positive rapid antigen test (RAT) for influenza A and/or influenza B (using a Sponsor-approved test kit), or positive test (using other methodology) for influenza A and/or B virus antigen or RNA performed in a clinical laboratory at the screening/enrollment evaluation are eligible for enrollment.

     OR
  2. Clinical Influenza with Negative Rapid Antigen Test (RAT). Subjects with a negative RAT test may be enrolled once the site has been approved by the Sponsor to enroll such subjects, based on documentation of an outbreak of influenza in the community. An influenza outbreak may be documented in the catchment area of the hospital via one of the following methods: 1) local confirmation of influenza A or B infection in the current influenza season by a) the institution's local laboratory, or b) the local public health system, or c) the national public health system, or d) a laboratory of a recognized multinational influenza surveillance scheme such as the European Influenza Surveillance Network (EISN); 2) prior enrollment of a RAT positive subject into this study at the same institution in the current influenza season.

     Exclusion Criteria:
* Subjects who have been hospitalized for greater than 24 hours (not including time spent in the Emergency Department).
* Treatment with any dose(s) of rimantadine, amantadine, ribavirin, zanamivir, or oseltamivir in the previous 7 days.
* Blood platelet count of < 20 x 109/L at the time of the screening evaluation.
* Serum bilirubin > 6 mg/dL or > 105 μmol/L at time of screening evaluation.
* Serum ALT or AST > 5 times the upper limit of normal at time of screening evaluation.
* Congestive heart failure of NYHA Class III or Class IV functional status.
* Serum creatinine > 5.0 mg/dL or > 500 μmol/L at time of screening evaluation.
* Subjects who require peritoneal dialysis.
* Altered neurologic status as defined by a Glasgow Coma Score of ≤ 9, unless medically induced.
* Females who are pregnant (positive urine or serum pregnancy test at screening evaluation) or breastfeeding.
* Actively undergoing systemic chemotherapy or radiotherapy treatment for a malignancy. Subjects who have completed treatment 30 days prior to enrollment are not excluded. Hormone treatment for cancer is also not excluded.
* Prior hematopoietic stem cell transplantation or solid organ transplant during the previous 4 months.
* HIV infection with a known CD4 count < 200 cells/mm3 unless on a stable highly active antiretroviral therapy (HAART) for at least 6 months.
* Presence of a pre-existing chronic infection that is undergoing or requiring medical therapy (eg, tuberculosis). Subjects with chronic osteomyelitis or Hepatitis B or C not requiring treatment are not excluded.
* Presence of any pre-existing illness that, in the opinion of the investigator, would place the subject at an unreasonably increased risk through participation in this study.
* Previous treatment with intravenous or intramuscular peramivir.
* Participation as a subject in any study of an experimental treatment for any condition within the 30 days prior to the time of the screening evaluation.
* Subjects diagnosed with Cystic Fibrosis.
* Subjects with confirmed clinical evidence of acute non-influenzal infection at the time of screening evaluation.
* Subjects who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (196):
- United States (60):
  - La Mesa, California
  - Long Beach, California
  - Modesto, California
  - Oceanside, California
  - Pulmonary Consultants PC Physicians Medical Group, Inc., Orange, California
  - Orange, California
  - UC Davis Medical Center, Sacramento, California
  - Sharp Chula Vista Medical Center, San Diego, California
  - San Diego, California
  - Denver, Colorado
  - Drogue Medical, LLC, Wheat Ridge, Colorado
  - Washington Hospital Center CAR, Washington D.C., District of Columbia
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Florida Hospital, Winter Park, Florida
  - Columbus, Georgia
  - DeKalb Medical Center, Decatur, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - Medical Arts Associates, Ltd., Moline, Illinois
  - Springfield, Illinois
  - South Bend, Indiana
  - Kentucky Lung Clinic, Hazard, Kentucky
  - Natchitoches, Louisiana
  - New Orleans, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University - Hutzel Hospital, Detroit, Michigan
  - Wayne State University, Department of Emergency Medicine, Detroit, Michigan
  - Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - Manhasset, New York
  - New York, New York
  - The Bronx, New York
  - University of North Carolina at Chapel Hill AIDS Clinical Trials Unit, Chapel Hill, North Carolina
  - Remington-Davis, Inc., Columbus, Ohio
  - Dayton, Ohio
  - Kettering, Ohio
  - Regional Infection Diseases Infusion Center Inc., Lima, Ohio
  - ID Clinical Research, LTD, Toledo, Ohio
  - Medical College Of Ohio, Toledo, Ohio
  - Toledo, Ohio
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - East Providence, Rhode Island
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Carilion Infectious Disease, Roanoke, Virginia
  - VA Medical Center - Salem, Salem, Virginia
- Argentina (9):
  - Hospital del Torax Dr. Antonio A. Cetrangolo, Buenos Aires
  - Buenos Aires
  - Caba
  - Córdoba
  - Mendoza
  - Merlo
  - Rosario
  - Santa Fe
  - Vicente López
- Belgium (3):
  - Brussels
  - Liège
  - Mons
- Bosnia and Herzegovina (2):
  - Sarajevo
  - Tuzla
- Brazil (9):
  - Belo Horizonte, Minas Gerais
  - Curitiba, Paraná
  - Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - Santo André, São Paulo
  - Santos, São Paulo
  - São Paulo, São Paulo
- Bulgaria (8):
  - Plovdiv
  - DDPPDI - Ruse, Rousse
  - Fifth MHAT-Sofia, AD, Sofia
  - MHAT - Tokuda Hospital Sofia, AD, Sofia
  - Military Medical Academy - MHAT, Sofia
  - Sofia
  - MHAT - Tokuda Hospital Sofia, AD, Stara Zagora
  - MHAT 'Dr. St. Cherkezov', AD, Veliko Tarnovo
- Canada (7):
  - Kelowna, British Columbia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- Chile (4):
  - Hospital Clinico Regional Dr. Guillermo Grant Benavente, Concepción
  - Hosp. de Urgencia Asistencia Publica Dr. Alejandro del Rio, Santiago
  - Santiago
  - Temuco
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Hradec Králové
  - Prague
  - Tábor
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Ustinad La, Ústí nad Labem
- Germany (6):
  - Berlin
  - Cologne
  - Erlangen
  - Göttingen
  - Mainz
  - Universitaetsklinikum Regensburg, Regensburg
- Hungary (5):
  - Debrecen
  - Fehérgyarmat
  - Principal SMO Dr. Bugyi Istvan Korhaz Szentes, Szentes
  - Fejer Megyei Szent Gyorgy Korhaz, Székesfehérvár
  - Zalaegerszeg
- India (28):
  - Hyderabad, Andhra Pradesh
  - Secunderabad, Andhra Pradesh
  - Ahmedabad, Gujarat
  - Karamsad, Gujarat
  - Surat, Gujarat
  - Vadodara, Gujarat
  - Faridabad, Haryana
  - Srinagar, Jammu and Kashmir
  - Bangalore, Karnataka
  - Mangalore, Karnataka
  - Ernākulam, Kerala
  - Thrissur, Kerala
  - Trivandrum, Kerala
  - Cherthala, Maharashtra
  - Mumbai, Maharashtra
  - Nagpur, Maharashtra
  - Nashik, Maharashtra
  - Pune, Maharashtra
  - Delhi, National Capital Territory of Delhi
  - Mohali, Punjab
  - Bikaner, Rajasthan
  - Fortis Escort Hospital, Jaipur, Rajasthan
  - Apollo First Med Hospitals, Chennai, Tamil Nadu
  - Life Line Multispecialty Hospital, Chennai, Tamil Nadu
  - Chennai, Tamil Nadu
  - Coimbatore, Tamil Nadu
  - Lucknow, Uttar Pradesh
  - Kolkata, West Bengal
- Israel (7):
  - Afula
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Ramat Gan
  - Tel Aviv
- Latvia (4):
  - Liepāja
  - Rēzekne
  - Valmiera
  - Ventspils
- Beirut, Lebanon
- Peru (3):
  - Arequipa
  - Cuzco
  - Lima
- Poland (6):
  - Bydgoszcz
  - Lodz
  - Mielec
  - Poznan
  - Puławy
  - Łańcut
- Russia (5):
  - Engel's
  - Niznhy Novgorod
  - Novosibirsk
  - Saint Petersburg
  - Tomsk
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Sad
- Trnava, Slovakia
- South Africa (10):
  - Middelburg, Mpumalanga
  - Bloemfontein
  - Dundee
  - Durban
  - Krugersdorp
  - Limpopo
  - Port Elizabeth
  - Pretoria
  - Somerset West
  - Worcester
- Ukraine (8):
  - Chernivtsi
  - Donetsk
  - Kharkiv
  - Kyiv
  - Odesa
  - Poltava
  - Sumy
  - Vinnytsia
- Leicester, United Kingdom

REFERENCES:
- [Derived] de Jong MD, Ison MG, Monto AS, Metev H, Clark C, O'Neil B, Elder J, McCullough A, Collis P, Sheridan WP. Evaluation of intravenous peramivir for treatment of influenza in hospitalized patients. Clin Infect Dis. 2014 Dec 15;59(12):e172-85. doi: 10.1093/cid/ciu632. Epub 2014 Aug 12. PMID 25115871

RESULTS

PARTICIPANT FLOW:
Groups:
- Peramivir+SOC: Adults (≥ 18 years): Peramivir (BCX-1812) 600 mg, administered intravenously, once daily (every 24 hrs) for 5 days (5 doses) in addition to institution's standard of care.
  Adolescents (12-17 years): Peramivir (BCX-1812) 10 mg/kg (not to exceed a maximum dose of 600 mg), administered intravenously, once daily (every 24 hrs) for 5 days (5 doses) in addition to institution's standard of care.
Period: Overall Study
Arm/Group | Placebo+SOC | Peramivir+SOC
Started | 137 | 268
Completed | 121 | 239
Not Completed | 16 | 29
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 2 | 6
Not completed — Withdrawal by Subject | 7 | 16
Not completed — Protocol Violation | 1 | 1
Not completed — Death | 2 | 1
Not completed — Noncompliance; Protocol Deviations | 2 | 3
Not completed — Missing | 1 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+SOC | Peramivir+SOC | Total
Number analyzed (Participants) | 137 | 268 | 405
Age, Continuous [Mean (Full Range); unit: years] | 43 [7 to 92] | 47 [6 to 92] | 46 [6 to 92]
Age, Customized [Number; unit: participants] — There were no subjects 6-11 years of age in the ITTI population.
  participants
    Children 6-11 Years | 2 | 2 | 4
    Adolescents 12-17 Years | 4 | 7 | 11
    Adults 18-24 Years | 23 | 33 | 56
    Adults 25-34 Years | 23 | 40 | 63
    Adults 35-44 Years | 21 | 44 | 65
    Adults 45-54 Years | 27 | 44 | 71
    Adults 55-64 Years | 17 | 45 | 62
    Adults 65-74 Years | 11 | 25 | 36
    Adults ≥ 75 Years | 9 | 28 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 132 | 199
  Male | 70 | 136 | 206
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 31 | 52 | 83
  White | 71 | 169 | 240
  Black, of African Heritage or African American | 23 | 28 | 51
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Other | 11 | 18 | 29
Body mass index (BMI) [Mean (Full Range); unit: kg/m^2] | 27.7 [15.2 to 59.9] | 27.5 [12.3 to 66.0] | 27.6 [12.3 to 66.0]
Supplemental oxygen required at Screening [Number; unit: participants]
  Needed | 45 | 87 | 132
  Not needed | 89 | 177 | 266
  Missing | 3 | 4 | 7
ICU admission at Baseline [Number; unit: participants]
  Admitted | 17 | 33 | 50
  Not admitted | 117 | 231 | 348
  Missing | 3 | 4 | 7
Influenza Vaccination Status [Number; unit: participants]
  Not vaccinated this year | 111 | 226 | 337
  Vaccinated this year | 26 | 41 | 67
  Missing | 0 | 1 | 1
Duration of Illness [Number; unit: participants]
  ≤ 48 hours | 75 | 150 | 225
  > 48 hours | 62 | 118 | 180
Standard of Care Received (CRF) [Number; unit: participants]
  NAI-Containing Antiviral Therapy | 89 | 179 | 268
  Non-NAI-Containing Antiviral Therapy | 9 | 7 | 16
  Supportive Care/No Antiviral Therapy | 39 | 82 | 121
Absolute Lymphocyte Count at Baseline [Mean (Standard Deviation); unit: cell count] | 1.3 (1.25) | 1.3 (1.52) | 1.3 (1.44)
Chest X-ray at Screening [Number; unit: participants]
  Normal | 88 | 148 | 236
  Abnormal | 49 | 120 | 169

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Resolution (Kaplan-Meier Estimate)
Description: Time to clinical resolution was defined as the time in hours from initiation of study treatment until normalization of at least 4 of the 5 signs within the respective normalization criteria, maintained for at least 24-hours. Time to clinical resolution was summarized by treatment group using the method of Kaplan-Meier. For subjects who did not experience clinical resolution, values were censored at the date of their last non-missing assessment of clinical resolution during the study (whether this assessment occurred as an inpatient or as an outpatient).
Time Frame: 10 days
Population: The Intent-to-Treat Infected-Non-NAI-Containing SOC (ITTI-Non-NAI) population included randomized subjects who received at least 1 dose of study drug, had confirmed influenza, and who received an SOC that does not contain a NAI at randomization.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 43 | 78
hours | 49.5 [40.0 to 61.9] | 42.5 [34.0 to 57.9]
Statistical Analysis 1: Comparison: Placebo+SOC vs Peramivir+SOC; Test type: Superiority or Other; p = 0.973, Wilcoxon-Gehan statistic; Analysis stratified by duration of illness at randomization, ICU status and use of supplemental oxygen at Baseline, influenza season and type; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.69 to 1.55] — The hazard ratio was calculated using a Cox regression model with factors of duration of illness at randomization, ICU status at Baseline, use of supplemental oxygen at Baseline, influenza season, and influenza type

2. Secondary Outcome: Change (Reduction) in Influenza Virus Titer
Description: The reduction in viral shedding was assessed as the change from baseline in log10 tissue culture infective dose50 (TCID50/mL) and RT-PCR and was summarized for each treatment group and study visit.
Time Frame: Baseline and 24, 48, 108 hours
Population: The Intent-to-Treat Infected-Non-NAI-Containing SOC (ITTI-Non-NAI) population included randomized subjects who received at least 1 dose of study drug, had confirmed influenza, and who received an SOC that does not contain an NAI at randomization.
Measure: Median (95% Confidence Interval); unit: log10 viral particles/mL
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 34 | 61
log10 viral particles/mL
  Change from Baseline, 24 Hours | -1.09 [-1.62 to -0.80] | -1.49 [-1.84 to -1.22]
  Change from Baseline, 48 Hours | -1.67 [-2.14 to -0.87] | -2.02 [-2.49 to -1.46]
  Change from Baseline, 108 Hours | -2.39 [-3.29 to -1.59] | -2.48 [-3.05 to -2.11]

3. Secondary Outcome: Time to Alleviation of Clinical Symptoms of Influenza
Description: Time to alleviation of clinical symptoms of influenza was measured as the time from the first dose of study drug through the time period in which all 7 symptoms of influenza (cough, sore throat, nasal congestion, myalgia [aches and pains], headache, feverishness, and fatigue) were absent or rated as no greater than mild for at least 24 hours. Time to alleviation of symptoms was estimated using the method of Kaplan-Meier. Subjects who did not have resolution of any individual clinical sign were censored at the time of their last non-missing assessment of that sign.
Time Frame: 10 days
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 43 | 77
hours | 68.2 [63.0 to 86.0] | 67.0 [59.0 to 78.8]
Statistical Analysis 1: Comparison: Placebo+SOC vs Peramivir+SOC; Test type: Superiority or Other; p = 0.558, Wilcoxon-Gehan statistic; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.75 to 1.72] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Resolution of Fever (Kaplan-Meier Estimate)
Description: Time to resolution of fever was measured as the time from initiation of study treatment until resolution of fever, maintained for at least 24 hours; temperature measurements taken less than 4 hours after antipyretic use were treated as missing values.
Time Frame: 10 days
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 43 | 78
hours | 41.0 [28.0 to 58.9] | 42.5 [32.0 to 56.4]
Statistical Analysis 1: Comparison: Placebo+SOC vs Peramivir+SOC; Test type: Superiority or Other; p = 0.633, Wilcoxon-Gehan statistic; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.59 to 1.31] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Resumption of Usual Activities
Description: Time to resumption of usual activities was determined from the visual analog scale (scale ranged from 0 to 10 where 0 indicated subject was unable to perform usual activities at all and 10 indicated subject was able to perform all usual activities fully). Time to resumption of usual activities was summarized by treatment group using the method of Kaplan-Meier.
Time Frame: 10 days
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 42 | 74
days | 9.3 [7.1 to 12.8] | 8.1 [5.1 to 9.3]
Statistical Analysis 1: Comparison: Placebo+SOC vs Peramivir+SOC; Test type: Superiority or Other; p = 0.747, Wilcoxon-Gehan statistic; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [0.92 to 2.32] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Subjects With ICU Admission
Description: The number of subjects requiring ICU admission post-randomization was summarized by treatment group.
Time Frame: 10 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 43 | 78
participants
  At Baseline | 8 | 15
  After initiation of treatment | 1 | 0
  At any time | 9 | 15

7. Secondary Outcome: Duration of All ICU Admissions (Kaplan-Meier Estimate)
Description: Duration of postbaseline ICU admission was defined as the total number of days in the ICU for those subjects who had a post-baseline admission to the ICU. Only days starting after the initial postbaseline admission were included. If a subject's stay in the ICU was ongoing, the duration was censored at the last study visit. Subjects who did not have a postbaseline admission had a duration of 0.
Time Frame: 10 days
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 43 | 78
days | 3.0 [2.0 to 6.0] | 3.0 [3.0 to 4.0]
Statistical Analysis 1: Comparison: Placebo+SOC vs Peramivir+SOC; Test type: Superiority or Other; p = 0.303, Wilcoxon-Gehan statistic; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.41 to 2.98] — The hazard ratio is calculated using a Cox regression model with factors of duration of illness at randomization, ICU status at baseline, use of supplemental oxygen at baseline, influenza season, and influenza type

8. Other Pre Specified Outcome: Time to Hospital Discharge
Description: Time to hospital discharge, defined as the number of days from initiation of study treatment until the subject was discharged from the hospital, was summarized by treatment group using the method of Kaplan-Meier. Subjects who were not discharged from the hospital were censored at their last study visit.
Time Frame: 10 days
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 43 | 78
days | 5.0 [5.0 to 6.0] | 5.0 [NA to NA] — The number of observed events was too small to allow estimation of the required parameter.

9. Other Pre Specified Outcome: Incidence of Influenza-Related Complications
Description: Influenza-related complications were defined as the occurrence of sinusitis, otitis, bronchitis, and pneumonia as reported on the influenza-related complications CRF.
Time Frame: 10 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 43 | 78
participants
  Any Influenza-Related Complication | 9 | 15
  Otitis | 0 | 0
  Sinusitis | 1 | 2
  Bronchitis | 4 | 5
  Pneumonia | 4 | 8
Statistical Analysis 1: Comparison: Placebo+SOC vs Peramivir+SOC; Test type: Superiority or Other; p = 0.768, Cochran-Mantel-Haenszel; Analysis stratified by symptom onset prior to randomization, Baseline ICU status, need for supplemental oxygen at Baseline, influenza season and type

10. Other Pre Specified Outcome: Number of Subjects Requiring More Than 5 Days of Study Drug
Description: Subjects who had not met the protocol-defined criteria of clinical resolution on Day 5 or who had detectable virus by RT-PCR from a sample collected on Study Day 4 after dosing continued their assigned treatment for a further 5 days.
Time Frame: 10 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 43 | 78
participants | 3 | 6
Statistical Analysis 1: Comparison: Placebo+SOC vs Peramivir+SOC; Test type: Superiority or Other; p = 0.758, Cochran-Mantel-Haenszel; [statistical method as in outcome 9, analysis 1]

11. Other Pre Specified Outcome: Survival at 14 and 28 Days After Initiation of Study Drug (Kaplan-Meier Estimate)
Description: Survival was calculated as the number of days from initiation of study drug until death or last contact. Estimates and 95% confidence intervals were calculated using the method of Kaplan-Meier and presented by treatment group.
Time Frame: 28 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent Survival
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 42 | 72
Percent Survival
  14 Day Survival | 98 [84 to 100] | 100 [100 to 100]
  28 Day Survival | 98 [84 to 100] | 100 [100 to 100]

12. Other Pre Specified Outcome: Initial Viral Sensitivity to Peramivir, Oseltamivir, and Zanamivir; IC50 (nM)
Description: Initial viral sensitivity to peramivir, oseltamivir, and zanamivir was assessed over time during the study, and was presented by influenza virus subtype. Initial assessment of susceptibility may have occurred at a post-baseline visit.
Time Frame: Initial (baseline or post-baseline) and up to 10 days
Population: The Intent-to-Treat Infected (ITTI) population included randomized subjects who received at least 1 dose of study drug, and had confirmed influenza A or B.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 116 | 222
nM
  A: H3N2-Initial Peramivir Susceptibility | 0.18 (0.074) | 0.18 (0.044)
  A: H3N2-Initial Oseltamivir Susceptibility | 0.30 (0.131) | 0.31 (0.131)
  A: H3N2-Initial Zanamivir Susceptibility | 0.34 (0.185) | 0.34 (0.071)
  A: H1N1- Initial Peramivir Susceptibility | 0.24 (0.152) | 1.11 (6.181)
  A: H1N1- Initial Oseltamivir Susceptibility | 1.12 (0.772) | 11.03 (70.524)
  A: H1N1- Initial Zanamivir Susceptibility | 0.60 (0.416) | 0.60 (0.402)
  B: Initial Peramivir Susceptibility | 1.14 (0.625) | 1.15 (0.628)
  B: Initial Oseltamivir Susceptibility | 18.47 (4.830) | 21.47 (9.422)
  B: Initial Zanamivir Susceptibility | 2.36 (1.009) | 2.30 (0.958)

13. Other Pre Specified Outcome: Change in Viral Sensitivity to Peramivir, Oseltamivir, and Zanamivir; Fold Change From Initial
Description: Viral sensitivity to peramivir, oseltamivir, and zanamivir was assessed over time during the study, and was presented as fold change from initial sensitivity by influenza virus subtype. Initial assessment of susceptibility may have occurred at a post-baseline visit.
Time Frame: Initial (baseline or post-baseline) and up to 10 days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Placebo+SOC | Peramivir+SOC
Number analyzed (Participants) | 116 | 222
fold change
  A: H3N2-Fold Change in Peramivir Susceptibility | 1.23 (0.555) | 1.19 (0.527)
  A: H3N2-Fold Change in Oseltamivir Susceptibility | 1.36 (0.836) | 1.14 (0.805)
  A: H3N2-Fold Change in Zanamivir Susceptibility | 2.70 (6.563) | 1.33 (0.773)
  A: H1N1-Fold Change in Peramivir Susceptibility | 1.12 (0.879) | 3.63 (16.333)
  A: H1N1-Fold Change in Oseltamivir Susceptibility | 1.51 (1.695) | 9.20 (50.920)
  A: H1N1-Fold Change in Zanamivir Susceptibility | 1.03 (0.728) | 1.06 (0.490)
  B: Fold Change in Peramivir Susceptibility | 1.01 (0.331) | 3.21 (8.456)
  B: Fold Change in Oseltamivir Susceptibility | 0.98 (0.376) | 1.48 (1.635)
  B: Fold Change in Zanamivir Susceptibility | 1.02 (0.375) | 1.36 (0.613)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded at least once daily during the period of study drug administration in the hospital and at each follow-up visit until the study completion visit at Day 14 or later.
Description: For subjects who experienced the same coded event more than once, only one event is presented. Seven of the 405 subjects who were randomized did not receive study drug; safety analyses included 398 subjects (134 in the Placebo+SOC arm and 264 in the Peramivir+SOC arm).
Arm/Group | Placebo+SOC | Peramivir+SOC
Serious Adverse Events (participants affected / at risk) | 13/134 | 15/264
Other Adverse Events (participants affected / at risk) | 42/134 | 63/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+SOC (N=134) | Peramivir+SOC (N=264)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Klebsiella Bacteraemia (Infections and infestations) | 0 | 1
Sinusitis Bacterial (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Echinococciasis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Viral Myositis (Infections and infestations) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 2
Neuroleptic Malignant Syndrome (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Multi-organ Disorder (General disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Accidental Needle Stick (Injury, poisoning and procedural complications) | 1 | 0
Haemodynamic Instability (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+SOC (N=134) | Peramivir+SOC (N=264)
Diarrhoea (Gastrointestinal disorders) | 10 | 12
Nausea (Gastrointestinal disorders) | 10 | 10
Constipation (Gastrointestinal disorders) | 7 | 6
Vomiting (Gastrointestinal disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 1 | 10
Anxiety (Psychiatric disorders) | 3 | 5
Alanine Aminotransferase Increased (Investigations) | 5 | 7
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 7
Aspartate Aminotransferase Increased (Investigations) | 3 | 6
Blood Glucose Increased (Investigations) | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1
Headache (Nervous system disorders) | 2 | 7
Dizziness (Nervous system disorders) | 3 | 1
Hypertension (Vascular disorders) | 1 | 7
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4

LIMITATIONS AND CAVEATS:
Interim analysis of the primary efficacy endpoint (time to clinical resolution) performed after the end of the 2012 Southern Hemisphere influenza season lead to study termination for futility. Final enrollment was ~70% of the planned enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No